CLINICAL TRIAL: NCT05393648
Title: Bipolar Efficacy Biomarkers for Accelerated Intermittent Theta Burst rTMS Trial
Brief Title: Bipolar Efficacy Biomarkers for rTMS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of Pennsylvania (Other); Milken Institute (Other)
Responsible Party: Principal Investigator, Itay Hadas, Assistant Research Scientist, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 800601
Record Dates: First submitted 2022-05-05; First posted 2022-05-26 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Bipolar Disorder; Bipolar Depression
Keywords: theta burst stimulation; accelerated TBS
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Patients enrolled in the study will be randomized to sham vs. active accelerated iTBS in a 1:1 ratio. Treatments will be over 1 week.
Who Masked: Participant, Outcomes Assessor
Masking Description: A sham component will be used over the right DLPFC for unilateral aiTBS treatment. This treatment component will mitigate concerns of expectancy, and will lead to blinding for patients. The Cool B65 A/P coil is unmarked, with one side producing active treatment and the other sham treatment with concurrent electrical stimulation, which accurately mimics active stimulation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active iTBS (Experimental): Patients will receive unilateral accelerated theta-burst stimulation to the left dorsal lateral prefrontal cortex for 5 consecutive days, with a total of 10 hours a day. Treatment will be 10min with 50min of breaks in between the 10 sessions.
  Interventions: Device: Accelerated Theta Burst Stimulation
- Sham iTBS (Placebo Comparator): Patients will receive sham unilateral accelerated theta-burst stimulation to the left dorsal lateral prefrontal cortex for 5 consecutive days, with a total of 10 hours a day. Treatment will be 10min with 50min of breaks in between the 10 sessions.
  Interventions: Device: Sham accelerated Theta Burst Stimulation

INTERVENTIONS:
Device: Accelerated Theta Burst Stimulation — Cool B65- A/P - active side magnetic coil stimulation applied to the left dorsal lateral prefrontal cortex.
  Arms: Active iTBS
Device: Sham accelerated Theta Burst Stimulation — Cool-B65 A/P - sham side magnetic coil stimulation applied to the left dorsal lateral prefrontal cortex.
  Arms: Sham iTBS

SUMMARY:
The research study is being conducted to test whether using high dose spaced theta-burst rTMS (a form of repetitive transcranial magnetic stimulation) produces a significant reduction in depressive symptoms compared with sham. This project will recruit patients aged 18-70 with symptoms of bipolar depression (BPD) who have failed (or not shown signs of improvement) after at least two prior treatments. The null hypothesis is that there will be no difference in reductions in depressive symptoms by the end of a five-day treatment period. The alternative hypothesis is that, compared with sham, active TMS will result in a greater reduction in depressive symptoms by the end of the treatment period.

To facilitate the development of rTMS protocols there is a need for biomarkers that are sensitive to BPD symptom severity and clinical improvement. Previously in our lab, investigators developed biomarkers suitable for depression trials, and these biomarkers are very likely to show sensitivity to BPD, since they are associated with brain regions and functions associated with BPD. As a secondary aim, the investigators will try to identify biomarkers in cortical region associated with BPD, and formulate a statistical model that may be able to predict BPD remission after the treatment. this study will lead to development of new brain stimulation treatment protocols and biomarkers, will aid in treatment selection, and eventually lead to better clinical outcome for patients suffering from BPD.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar depression (BP I and BP II) by DSM 5 criteria (Diagnostic and Statistical Manual of Mental Disorders, 2013)
* Age 18-70
* Right or left handed
* All genders
* Treatment resistant depression, as in they must have treatment resistant depression with 2 or more prior antidepressant trials that have failed to produce a response (> 50% reduction in symptoms) using ATHF criteria (Sackeim et al., 2019)
* Able to provide informed consent to participate in the study
* Must be on a stable medication regimen, requiring at least one mood stabilizer
* Depression severity as represented by scoring at least 20 on MADRS
* Meet the safety criteria as defined in the transcranial magnetic stimulation adult safety screen (TASS).

Exclusion Criteria:

* No current substance abuse disorder for the past 6 months (previous substance abuse not exclusionary)
* Any psychotic disorder or current active psychotic symptoms (personality disorders not exclusionary unless in the opinion of the referring psychiatrist it would jeopardize participation)
* No dementia or other major neurological disorders
* Not having depression as primary disorder
* No major medical illness, for example metastatic cancer, end stage renal disease
* Not able to verify contact information. Participants must be able to follow through with the study & must have verified contact information and at least one verified contact
* Pregnancy. While there are no known risks to a fetus this is a new use of TMS, which has not been tested, thus pregnancy is exclusionary
* Score on YMRS greater than 12 (patients with mixed features have been shown not to respond well to TMS treatment (Tavares et al., 2021).
* Rapid cycling Bipolar illness (patients with > 4 mood episodes within the past year will be excluded, as they have a higher risk of switch to mania (Tondo et al., 2010)
* Any implants, conditions, or contraindications that would be deemed unsafe for TMS or MRI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) Scores | 6 months
  Assessment of the clinical efficacy, safety, and tolerability of aiTBS for depressive symptoms in BPD by analysis of scores on the Montgomery-Asberg Depression Rating Scale (MADRS) obtained at baseline, post-treatment, and throughout the course of treatment, and comparing them between active vs. sham TMS treatment groups. Scores on the MADRS range from 0 to 60, with higher scores indicating more severe depression.
Change in Hamilton Rating Scale for Depression (HRSD-17) Scores | 6 months
  Assessment of the clinical efficacy, safety, and tolerability of aiTBS for depressive symptoms in BPD by analysis of scores on the Hamilton Rating Scale for Depression (HRSD-17) obtained at baseline, post-treatment, and throughout the course of treatment, and comparing them between active vs. sham TMS treatment groups. Scores on the MADRS range from 0 to 53, with higher scores indicating more severe depression.
Assessment of Biomarkers | 6 months
  Analysis of transcranial magnetic stimulation concurrent with electroencephalogram (TMS-EEG) to extract effective connectivity metrics between the subgenual cingulate (SGC) and the left dorsolateral prefrontal cortex (DLPFC) as BPD biomarkers, as measured by scores on the HAMD and MADRS, for aiTBS compared to sham treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Interventional Psychiatry, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No